CLINICAL TRIAL: NCT06751147
Title: Effects of Lateral Femoral Cutaneous Nerve Mobilization With and Without Muscle Energy Techniques on Neuropathic Pain, Knee Range of Motion and Quality of Life in Pregnant Females
Brief Title: Effects of Lateral Femoral Cutaneous Nerve Mobilization With and Without Muscle Energy Techniques in Pregnant Females
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/00234 Mehwish
Record Dates: First submitted 2024-12-20; First posted 2024-12-27 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Meralgia Paresthetica
Keywords: femoral neuropathy
MeSH Terms: conditions — Femoral Neuropathy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: outcome assessor was kept blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Experimental): Lateral Femoral cutaneous nerve mobilization with muscle energy techniques
  Interventions: Other: Group A
- GROUP B (Experimental)
  Interventions: Other: Experimental Group B

INTERVENTIONS:
Other: Group A — It consists of 24 patients who were assessed by prone knee bend (PKB) test and knee range of motion was measured by goniometer. In addition to traditional physical therapy and muscle energy procedures, patients in this group received neural mobilization. The patient laid on their side with their knee bent to a 90-degree angle and the affected side looking up while neural mobilization was carried out. The therapist then performed the technique by abducting and extending the patient's hip. Five repetitions of the nerve stretch were performed, each with a 10-second hold and a 5-second rest in between.
  METs were implemented in two positions using post-isometric relaxation (PIR): In this initial posture, the patient laid on their back with the affected leg just over the bed's edge. With one hand, the physiotherapist stood facing the affected side and pressed the contralateral ASIS to keep the patient from rolling off the bed. The therapist, however, simultaneously grabbed the femur dist
  Arms: group A
Other: Experimental Group B — It involves 24 patients who had received the neural mobilization described above along with traditional physical therapy that does not involve muscular energy techniques. The treatment took place in the outpatient physical therapy department and lasted around thirty minutes in total
  Arms: GROUP B

SUMMARY:
The rationale of this study is to provide empirical evidence regarding the efficacy and safety of neural mobilization in pregnant women with meralgia paresthetica. By investigating the potential benefits of this intervention, healthcare professionals can make informed decisions about incorporating neural mobilization into the management of this condition during pregnancy. Focusing on the impact of neural mobilization and muscle energy techniques on both neuropathic pain and quality of life aligns with a patient-centered approach to care. The goal is not only to reduce symptoms but also to enhance overall well-being and functional capacity

DETAILED DESCRIPTION:
The literature gap of the study is that upto our knowledge, there is little or no evidence found in previous researches on the combined effects of lateral femoral cutaneous nerve mobilization in combination with MET in pregnant females. Secondly no quantitative measurement as range of motion with goniometer has been yet studied

ELIGIBILITY:
Inclusion Criteria:

* Age ranges from 18 to 40 years
* Body mass index ≥25kg/m2.
* Pregnant females in third trimester diagnosed with myalgia paraesthetica.
* Multigravida pregnant females
* Patients will be screened through Prone Knee Bend (PKB) test for femoral nerve compression.
* Positive pelvic compression test(1)

Exclusion Criteria:

* Those having other entrapment syndromes or radicular symptoms
* Motor weakness
* Having a history or ongoing cancerous proliferation
* Active infection

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — patients are of Pregnant females
Enrollment: 48 (Actual)
Dates: Start 2024-12-23 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2025-05-15 (Actual)

PRIMARY OUTCOMES:
quality of life is assessed by QOL questioner | at base line pre intervention, at the end of 4th week post intervention
  EQ-5D is used to measure quality of life
Knee range of motion is used to measure ROM | at base line pre intervention, at the end of 4th week post intervention
  measured by goniometer
neuropathic pain | at base line pre intervention, at the end of 4th week post intervention
  The Neuropathic Pain Scale (NPS) is a tool used to assess the specific qualities of pain associated with neuropathic pain. It helps differentiate neuropathic pain from other types of pain by evaluating different pain sensations and their intensity. The NPS consists of 10 items, each rated on a scale of 0 to 10, where 0 is "no pain" and 10 is the "worst imaginable pain".

CONTACTS AND LOCATIONS:
Overall Officials: Iqra abdul ghafoor, PPDPT, Principal Investigator — Riphah International University
Locations (2):
- Pakistan (2):
  - Ghurkhi Hospital, Lahore, Punjab Province
  - Ghurki Hospital, Lahore, Punjab Province

IPD SHARING:
Plan to Share IPD: No